CLINICAL TRIAL: NCT06889714
Title: Investigation of the Effects of Frailty and Sarcopenia on Postoperative Recovery and Complications in Geriatric Patients Undergoing Colorectal Cancer Surgery
Brief Title: Investigation of the Effects of Frailty and Sarcopenia on Postoperative Recovery and Complications in Geriatric Patients
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ferda YAMAN, Associate Professor, Eskisehir Osmangazi University
Other Study IDs: Eskisehir
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Frailty; Sarcopenia
Keywords: geriatric anesthesia; sarcopenia; ultrasonography; postoperative complications; quadriceps femoris
MeSH Terms: conditions — Frailty; Sarcopenia; Postoperative Complications | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasonography — Right thigh length (between the right femur greater trochanter and patella) was measured and recorded while the patients were lying supine. A linear transducer (Philips Affiniti 50, Philips Medical Systems, Seattle, WA, United States) was used for ultrasonographic measurements. The rectus femoris (RF) and vastus intermedius (VI) were visualized with the feather-touch technique after a generous amount of ultrasound gel was sprayed in the center of the right thigh, and the thickness of the muscles was determined and recorded using ultrasonography software. After these measurements, the rectus femoris-to-thigh length ratio (RF/B), vastus intermedius-to-thigh length ratio (VI/B), and total muscle thickness-to-thigh length ratio (T/B) were calculated and recorded.

SUMMARY:
After obtaining ethical approval, 42 patients with American Society of Anesthesiologists (ASA) scores I-III who were scheduled for surgery under general anesthesia were included in our prospective study. Patients were monitored in the preoperative preparation room in the operating room and frailty was assessed using the FRAIL scale and sarcopenia was assessed using the STAR ratio. The thickness of the rectus femoris and vastus intermedius muscles of the patients was measured and recorded by ultrasonography. Thigh lengths were measured and recorded. Rectus Femoris/Thigh Length (RF/B), Vastus Intermedius/Thigh Length (VI/B), and Total Muscle Thickness/Thigh Length (T/B) were calculated and recorded. Patients were followed up according to the Modified Aldrete Score after surgery in the anesthesia recovery unit, and the time to reach 9-10 points was recorded, and the time to leave the recovery unit was recorded. Postoperatively, complications were followed up according to the Clavien-Dindo Classification, and discharge times from the hospital were recorded.

DETAILED DESCRIPTION:
Frailty is a clinically identifiable state of heightened vulnerability resulting from age-related declines in physiological systems and functions, leading to impaired resilience to stressors. Frailty is highly prevalent among the elderly and is associated with an increased risk of falls, disability, hospitalization, and mortality. Magnetic resonance imaging (MRI) and computed tomography (CT) are considered the gold standard for sarcopenia diagnosisCT is also limited due to radiation exposure and similar logistical constraints. In contrast, ultrasonography (USG) is portable, cost-effective, and can be performed at the bedside without radiation exposure.

Using high-frequency ultrasound probes, peripheral muscle tissues and their dimensions can be rapidly assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients over 60 years of age who are undergoing colorectal malignancy surgery under general anesthesia
* patients willing to participate in the study
* Patients with ASA score I-III

Exclusion Criteria:

* Patients with Parkinson's disease,
* Alzheimer's disease,
* history of cerebrovascular events,
* neuromuscular disease,
* cognitive dysfunction,
* severe liver disease,
* severe heart disease,
* impaired cooperation due to kidney disease,
* emergency and trauma patients,
* patients with bilateral lower extremity amputations

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — all genders were accepted to the study without gender discrimination
Study Population: 42 patients over 60 years of age with ASA score I-III who were to undergo colorectal malignancy surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
age | 1 year
  years old
sex | 1 year
  female, male
height | 1 year
  meter
body weight | 1. year
  kg
educational status | 1 year
  primary school graduate, middle school graduate, high school graduate, university graduate
marital status | 1 year
  married, single, widowed
ASA score | 1 year
  American Society of Anesthesiologists' Classification (ASA 1,2,3,4,5)
rectus femoris muscle thickness | 1 year
  cm
vastus intermedius(VI) thickness | 1 year
  cm
rectus femoris-to-thigh length ratio | 1 year
  ratio
vastus intermedius-thigh length ratio | 1 year
  ratio
total muscle thickness to thigh length ratio | 1 year
  ratio
frailty score | 1 year
  0-NORMAL, 1-2 PRE-FRAİL, 3-5 FRAİL
recovery time from anesthesia | 1 year
  minutes
hospital discharge time | 1 year
  days
Modified Clavien-Dindo Classification | 1 year
  1, 2, 3A, 3B, 4A, 4B, 5

CONTACTS AND LOCATIONS:
Overall Officials: ferda yaman, Assoc prof, Principal Investigator — University of Eskişehir Osmangazi
Locations (1):
- University of Eskisehir Osmangazi, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No